CLINICAL TRIAL: NCT02062047
Title: Full-mouth and Partial-mouth Scaling and Root Planing in Type 2 Diabetic Subjects: Clinical, Immunological and Microbiological Outcomes
Brief Title: Full-mouth and Partial-mouth Scaling and Root Planing in Type 2 Diabetic Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Guarulhos (Other)
Responsible Party: Principal Investigator, Poliana Mendes Duarte, PhD, University of Guarulhos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SISNEP/277
Record Dates: First submitted 2014-02-07; First posted 2014-02-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Periodontitis; Diabetes
Keywords: Diabetes Mellitus; Chronic Periodontitis; Root Planing; Cytokines; microbiology; Glycated hemoglobin; diabetic subjects
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus; Chronic Periodontitis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FMSRP+CLX (Experimental): Full-mouth scaling and root planing in a maximum of 24 hours, application and irrigation of chlorhexidine 2% gel, rinsing chlorhexidine 0.12% solution during 60 days
  Interventions: Procedure: FMSRP; Drug: Chlorhexidine
- FMSRP + placebo group (Placebo Comparator): Full-mouth scaling and root planing in a maximum of 24 hours, application and irrigation of placebo, rinsing placebo solution during 60 days
  Interventions: Procedure: FMSRP; Other: Placebo
- PMSRP group (Active Comparator): Partial-mouth scaling and root planing in 4-6 sessions in a maximum of 2 weeks
  Interventions: Procedure: PMSRP

INTERVENTIONS:
Procedure: FMSRP — FMSRP in a maximum of 24 hours.
  Arms: FMSRP + placebo group; FMSRP+CLX
Drug: Chlorhexidine — Application and irrigation of chlorhexidine, rinsing chlorhexidine solution during 60 days
  Other Names: (N/A)
  Arms: FMSRP+CLX
Procedure: PMSRP — Scaling and root planing in 4-6 sessions in a maximum of 2 weeks
  Arms: PMSRP group
Other: Placebo — Application and irrigation of placebo, rinsing placebo solution during 60 days
  Arms: FMSRP + placebo group

SUMMARY:
The aim of this study will be to evaluate: 1- the effect of full-mouth (FM) scaling and root (SRP) planing in 24 hours associated with or without extensive application of chlorhexidine (CLX) on clinical, microbiological, glycemic and immunological parameters in diabetic subjects with chronic periodontitis at 3, 6 and 12 months post-therapy. The hypothesis is that FMSRP associated with CLX use will provide the best clinical, microbiological, glycemic and immunological outcomes for the treatment of diabetic subjects with periodontitis. Sixty diabetic subjects with chronic periodontitis will be divided in the following therapeutic groups (n=20 subjects per group): FMSRP+CLX group - FMSRP in a maximum of 24 hours, application and irrigation of chlorhexidine 2% gel, rinsing chlorhexidine 0.12% solution during 60 days; FMSRP + placebo group - FMSRP in a maximum of 24 hours, application and irrigation of placebo, rinsing placebo solution during 60 days; Partial-mouth (PM) SRP group: SRP in 4-6 sessions in a maximum of 2 weeks. The following clinical parameters will be evaluated at 3, 6 and 12 months post-therapy: plaque accumulation, gingival bleeding, probing depth, clinical attachment level, bleeding on probing and suppuration. At these same periods, glycated hemoglobin levels will be obtained from all subjects. In addition, six subgingival biofilm samples per subject will be analyzed by checkerboard DNA-DNA hybridization for 40 bacterial species at baseline, 3, 6 and 12 post-therapy. Finally, gingival crevicular fluid samples from two shallow and two deep sites will be evaluated for the levels of cyto/chemokines by ELISA. Data will be submitted to appropriate statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes mellitus
* Clinical diagnosis of generalized chronic periodontitis
* > 30 years old
* At least 15 teeth excluding third molars and teeth indicated to exodontia
* More than 30% of the sites with probing depth and clinical attachment level ≥ 4 mm at baseline

Exclusion Criteria:

* Pregnancy
* Lactation
* Current smoking
* Smoking within the past 5 years
* Periodontal or/and antibiotic therapies in the previous 6 months
* Regular use of mouthrinses containing antimicrobials in the preceding 2 months
* Other systemic condition that could affect the progression of periodontal disease
* Long-term use of anti-inflammatory and immunosuppressive medications
* Presence of periapical pathology
* Use of orthodontic appliances
* Multiple systemic complications of DM.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Changes in clinical attachment level (CAL) in sites with initial PD ≥7mm from baseline to 12 months. | From baseline to 12 months

SECONDARY OUTCOMES:
Changes in percentage of sites with probing depth ≥5mm | From baseline to 12 months
Changes in serum levels of glycemic hemoglobin | From baseline to 12 months
Changes in the counts of pathogenic bacterial species | From baseline to 12 months
Changes in the levels of tumor necrosis factor-α in gingival crevicular fluid | From baseline to 12 months
Changes in the levels of plaque accumulation | From baseline to 12 months
Changes in the mean percentage of sites with bleeding on probing | From baseline to 12 months
Changes in the full-mouth probing depth | From baseline to 12 months
Changes in the serum levels of fasting plasma glucose | From baseline to 12 months
Changes in the proportions of pathogenic bacterial species | From baseline to 12 months
Changes in the levels of interferon (IFN)-γ in gingival crevicular fluid | From baseline to 12 months
Changes in the levels of interleukin (IL)-17 in gingival crevicular fluid | From baseline to 12 months
Changes in the levels of IL-23 in gingival crevicular fluid | From baseline to 12 months
Changes in the levels of IL-4 in gingival crevicular fluid | From baseline to 12 months
Changes in levels of receptor activator of NF-κß ligand (RANKL) in gingival crevicular fluid | From baseline to 12 months
Changes in the levels of osteoprotegerin (OPG) in gingival crevicular fluid | From baseline to 12 months